CLINICAL TRIAL: NCT02206412
Title: Role of High Mobility Group Box 1 as a Prognostic Biomarker in Patients Undergoing Off-pump Coronary Artery Bypass Graft
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0341
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2014-07

CONDITIONS: Coronary Artery Occlusive Disease
Keywords: high mobility group box 1; prognostic biomarker; off-pump coronary artery bypass graft; patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HMGB1 group

SUMMARY:
High mobility group 1 (HMGB1) protein is both a nuclear factor and a secreted protein, and has recently been identified as a cytokine mediator of systemic inflammation. HMGB1 is released by inflammatory cells actively, or increased during cell death passively and mediates inflammatory response. It has been reported to have association with the prognosis after acute coronary syndrome, ischemia-reperfusion injury of myocardium, atherosclerosis and heart failure. This study aimed to investigate the relationship of serum levels of HMGB1 and post operative prognosis of patients who had undergone off-pump coronary artery bypass graft.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20
2. Patients undergoing off-pump coronary artery bypass graft

Exclusion Criteria:

1. Age < 20
2. Patients undergoing off-pump coronary artery bypass graft with other simultaneous surgery
3. Patients participating other study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over age 20 who are undergoing off-pump coronary artery bypass graft
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2014-07; Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Maximum value of HMGB1 | Change from induction of anesthesia to 2hrs after transfer to intensive care unit
  Measure the maximum value of HMGB1 in all patients and calculate median value. And device into upper median value group and under median value group and compare frequency of composite morbidity/mortality rate between two groups. composite morbidity/mortality is as follows:
  1. Stroke
  2. Renal failure
  3. Prolonged ventilation more than 24 hours
  4. Deep sternal wound infection
  5. Reoperation for any reason
  6. Mortality during the hospitalization for surgery, even if over 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology & Pain Medicine, Yonsei university college of medicine, Seoul, South Korea